CLINICAL TRIAL: NCT06561425
Title: A Phase I/II, Multicenter Study Evaluating the Feasibility, Safety, and Efficacy of Point-of-care Manufactured GLPG5101 (19CP02) in Subjects With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Brief Title: A Study Evaluating the Safety and Efficacy of GLPG5101 (19CP02) in Participants With Non-Hodgkin Lymphoma
Acronym: Atalanta-1
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP0201-NHL; 2022-502661-23-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Relapsed/Refractory B-cell Non-Hodgkin Lymphoma; Lymphomas Non-Hodgkin&Amp;Amp;#39;s B-Cell
Keywords: non-Hodgkin lymphoma (NHL); Follicular lymphoma (FL); Marginal zone lymphoma (MZL); Mantle cell lymphoma (MCL); Burkitt lymphoma (BL); Primary central nervous system lymphoma (PCNSL); Diffuse large B-cell lymphoma (DLBCL); CAR T-cell therapy; Diffuse large B-cell lymphoma - Richter Transformation (DLBCL-RT); small lymphocytic leukemia (SLL); chronic lymphocytic leukemia (CLL)
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Phase 1 (Dose escalation phase): Dose level 1 (Experimental): Participants will receive a single dose of GLPG5101 intravenous (IV) cell suspension for infusion at dose level 1 on Day 0.
  Interventions: Genetic: GLPG5101
- Phase 1 (Dose escalation phase): Dose level 2 (Experimental): Participants will receive a single dose of GLPG5101 IV cell suspension for infusion at dose level 2 on Day 0.
  Interventions: Genetic: GLPG5101
- Phase 1 (Dose escalation phase): Dose level 3 (Experimental): Participants will receive a single dose of GLPG5101 IV cell suspension for infusion at dose level 3 on Day 0.
  Interventions: Genetic: GLPG5101
- Phase 2 (Dose expansion phase): Cohort 1a: DLBCL 2L+ (Experimental): Participants in this cohort will receive a single dose of GLPG5101 IV cell suspension for infusion at the selected RP2D level for this disease subtype on Day 0
  Interventions: Genetic: GLPG5101
- Phase 2 (Dose expansion phase): Cohort 1b: DLBCL 2L+ SCNSL (Experimental): Participants in this cohort will receive a single dose of GLPG5101 IV cell suspension for infusion at the selected RP2D level for this disease subtype on Day 0
  Interventions: Genetic: GLPG5101
- Phase 2 (Dose expansion phase): Cohort 2: High-risk first-line DLBCL (Experimental): Participants in this cohort will receive a single dose of GLPG5101 IV cell suspension for infusion at the selected RP2D level for this disease subtype on Day 0
  Interventions: Genetic: GLPG5101
- Phase 2 (Dose expansion phase): Cohort 3: Indolent B-cell NHL (FL and MZL 3L+) (Experimental): Participants in this cohort will receive a single dose of GLPG5101 IV cell suspension for infusion at the selected RP2D level for this disease subtype on Day 0
  Interventions: Genetic: GLPG5101
- Phase 2 (Dose expansion phase): Cohort 4: MCL 2L+ (Experimental): Participants in this cohort will receive a single dose of GLPG5101 IV cell suspension for infusion at the selected RP2D level for this disease subtype on Day 0
  Interventions: Genetic: GLPG5101
- Phase 2 (Dose expansion phase): Cohort 5: BL 2L+ (Experimental): Participants in this cohort will receive a single dose of GLPG5101 IV cell suspension for infusion at the selected RP2D level for this disease subtype on Day 0
  Interventions: Genetic: GLPG5101
- Phase 2 (Dose expansion phase): Cohort 6a: PCNSL 2L+ (Experimental): Participants in this cohort will receive a single dose of GLPG5101 IV cell suspension for infusion at the selected RP2D level for this disease subtype on Day 0
  Interventions: Genetic: GLPG5101
- Phase 2 (Dose expansion phase): Cohort 6b: PCNSL first-line consolidation (Experimental): Participants in this cohort will receive a single dose of GLPG5101 IV cell suspension for infusion at the selected RP2D level for this disease subtype on Day 0
  Interventions: Genetic: GLPG5101
- Phase 2 (Dose expansion phase): Cohort 7: DLBCL-RT 2L+ (Experimental): Participants in this cohort will receive a single dose of GLPG5101 IV cell suspension for infusion at the selected RP2D level for this disease subtype on Day 0
  Interventions: Genetic: GLPG5101
- Experimental: Phase 2 (Dose expansion phase): Cohort 8 CLL/SLL (r/r) (Experimental): Participants in this cohort will receive a single dose of GLPG5101 IV cell suspension for infusion at the selected RP2D level for this disease subtype on Day 0
  Interventions: Genetic: GLPG5101

INTERVENTIONS:
Genetic: GLPG5101 — Autologous anti-CD19 chimeric antigen receptor (CAR) T cell therapy
  Other Names: 19CP02

SUMMARY:
This study is evaluating whether an experimental treatment called GLPG5101 helps to treat non-Hodgkin lymphoma (NHL) and if it is safe to use.

This study will be carried out in 2 phases:

* The first phase is to see which doses of GLPG5101 work best with the least number of side effects.
* In the second phase, participants will receive the selected dose(s) based on the results in the first phase.

DETAILED DESCRIPTION:
Phase 1 Dose escalation phase:

The dose escalation phase is designed to select the doses for dose expansion based on efficacy and safety outcomes.

Three dose levels of GLPG5101 will be evaluated to determine the recommended phase 2 doses (RP2Ds).

Participants with aggressive or indolent forms of Relapsed/Refractory B-cell Non-Hodgkin Lymphoma (r/r NHL) including follicular lymphoma (FL), marginal zone lymphoma (MZL), mantle cell lymphoma (MCL), and Diffuse large B-cell lymphoma (DLBCL) will be enrolled. In case any safety or efficacy differences based on histological subtype of the disease are observed, it may be decided to make decisions regarding dose escalation for a specific subtype(s) independently, upon recommendation by the Safety Review Committee (SRC). Hence the RP2Ds may be different for different subtypes.

Phase 2 Dose expansion phase:

After determination of the RP2Ds, the study continues with the dose expansion phase. Different doses deemed safe by the SRC within the same indication may be explored in the dose-expansion phase to help select the optimal dose for further development.

During this phase, participants will be enrolled into separate disease cohorts as defined by their NHL subtype:

* Cohort 1a: DLBCL second line or greater (2L+)
* Cohort 1b: DLBCL 2L+ with secondary central nervous system lymphoma (SCNSL)
* Cohort 2: High-risk first-line DLBCL
* Cohort 3: Indolent B-cell NHL (FL and MZL third-line or greater [3L+])
* Cohort 4: MCL 2L+
* Cohort 5: BL 2L+
* Cohort 6a: PCNSL 2L+
* Cohort 6b: PCNSL first-line consolidation
* Cohort 7: DLBCL-RT 2L+
* Cohort 8: CLL/SLL (r/r)

Participants per disease cohort will be treated at the selected RP2Ds for that disease subtype.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of one of the following NHL subtypes: DLBCL, FL grade 1, 2 or 3A, MZL, MCL, BL, PCNSL, DLBCL-RT, High Grade B-cell Lymphoma (HGBL), CLL/SLL
* Relapsed or refractory disease
* Presence of at least one measurable lesion according to the Lugano classification (except for PCNSL subjects ineligible for ASCT after induction therapy, Cohort 6b; and except for CLL/SLL subjects without a measurable lesion or a PET positive lesion will be eligible if they have splenomegaly (spleen size >13 cm) and bone marrow infiltration with lymphoma)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (Participants with ECOG 2 must have serum albumin ≥ 3.4 gram/deciliter)
* Adequate bone marrow function
* Adequate renal, hepatic and pulmonary function
* Women of childbearing potential must have a negative serum pregnancy test at screening and prior to the first dose of conditioning chemotherapy
* Women of childbearing potential and all male subjects must agree to use highly effective methods of contraception and agree to remain on a highly effective method of contraception from the time of signing the informed consent form until at least 12 months after GLPG5101 infusion. Subjects must agree to not donate eggs or sperm during this period.

Key Exclusion Criteria:

* Selected prior treatments as defined in the protocol
* History of another primary malignancy that requires intervention beyond surveillance or that has not been in remission for at least 3 years. (exceptions per protocol)
* Toxicity from previous anticancer therapy that has not resolved to baseline levels or to ≤ Grade 2
* Active central nervous system (CNS) involvement (lesion on contrast-enhanced CT/MRI brain, malignant B cells in CSF) by disease under study (exceptions per protocol)
* Clinically significant cardiac disease
* Primary immunodeficiency
* Stroke or seizure within 6 months of screening
* History of autoimmune disease requiring systemic immunosuppression or disease modifying treatment within 28 days before screening
* Infection with human immunodeficiency virus (HIV), active hepatitis B or active hepatitis C virus
* Systemic fungal, bacterial, viral, or other infection that is not controlled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | 2 years
Phase 1: Number of participants with Dose-Limiting Toxicities (DLTs) | From first dose up to Day 28
Phase 2: Number of participants with objective response (OR) per the Lugano Classification or International Primary central nervous system lymphoma Collaborative Group (IPCG) criteria for PCNSL or per iwCLL (CLL [Cohort 8] and DLBCL-RT [Cohort 7] only) | 2 years
  For all cohorts

SECONDARY OUTCOMES:
Phase 2: Number of participants with AEs and SAEs | 2 years
Number of participants with AEs of special interests | 2 years
Number of participants with OR per the Lugano Classification or IPCG criteria | 2 years
  For phase 1 and cohort 6b only
Number of participants with OR per International workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria (DLBCL-RT [cohort 7] only | 2 years
Number of participants with complete response (CR) per Lugano Classification or IPCG criteria for PCNSL or per iwCLL (CLL [Cohort 8] and DLBCL-RT [Cohort 7] only) | 2 years
Duration of response (DOR) | 2 years
Duration of complete response (DOCR) | 2 years
Progression-free survival (PFS) | 2 years
Overall survival (OS) | 2 years
Number of participants without minimal Residual Disease (MRD) at CR (DLBCL, MCL, DLBCL-RT, and CLL/SLL) | 2 years
Pharmacokinetics (PK): Levels of anti-CD19 CAR T cells in blood at peak and over time | 2 years
Pharmacodynamics (PD): Levels of chemokines in serum over time | Day 7 before infusion, Day 0, Day 1, Day 4, Day 7, Day 10, Day 14, Day 21, Day 28
PD: Levels of cytokines in serum over time | Day 7 before infusion, Day 0, Day 1, Day 4, Day 7, Day 10, Day 14, Day 21, Day 28
Percentage of successfully manufactured GLPG5101 products within the predefined release specifications | From leukapheresis to infusion
Phase 2: Change from baseline in measurement of HRQoL using the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 and its CLL-specific module QLQ-CLL-17 (DLBCL-RT and CLL only), and EuroQol EQ-5D-5L | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (10):
- United States (3):
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
- Belgium (4):
  - Antwerp University Hospital, Edegem
  - UZ Leuven, Leuven
  - CHU De Liège, Liège
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - Leiden University Medical Center, Leiden
  - Erasmus Universitair Medisch Centrum Rotterdam (Erasmus MC), Rotterdam

IPD SHARING:
Plan to Share IPD: No